CLINICAL TRIAL: NCT02645149
Title: Molecular Profiling and Matched Targeted Therapy for Patients With Unresectable Advanced or Metastatic Melanoma
Acronym: Match Mel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melanoma Institute Australia (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIA2015/174
Record Dates: First submitted 2015-12-27; First posted 2016-01-01 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Melanoma
Keywords: Metastatic Melanoma; Molecular Testing; Targeted Therapy
MeSH Terms: conditions — Melanoma | interventions — Standard of Care; Clinical Trials as Topic; Immunotherapy; Biological Factors; trametinib; Palliative Care; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- A1. Non-V600 BRAF, BRAF wildtype, NRAS wildtype. Actionable gene mutation, matched drug available (Experimental): Patients will receive targeted drug matched to the actionable gene mutation detected on NGS testing. If a patient cannot receive the matched targeted therapy because of the existence of one or more drug specific exclusion criteria, an alternative matched therapy may be assigned, or trametinib, or clinical trials if available.
  Interventions: Drug: Matched targeted therapy
- A2. Non-V600 BRAF, BRAF wildtype, NRAS wildtype. Actionable gene mutation, no matched drug available (Experimental): Patients may have an actionable aberration for which there is no current study-specific drug supply available. In this scenario, access will be sought for compassionate use of the relevant approved targeted therapy.
  Interventions: Drug: Compassionate Access Targeted Therapy
- A3. Non-V600 BRAF, BRAF wild type and NRAS wild type melanoma - no actionable genetic aberration (Experimental): Patients for whom there is no actionable genetic aberration will receive trametinib, based upon the known MAPK excess activity in the majority of melanomas that may be inhibited by a MEK inhibitor
  Interventions: Drug: Trametinib and / or supportive care
- B. Mucosal melanoma (Experimental): Patients will receive combined trametinib and ribociclib based on evidence to suggest that combined MEK inhibition and CDK4/6 inhibition may be effective. After failure of trametinib and ribociclib, actionable genetic aberrations from the NGS testing will be reviewed for the opportunity to use a further targeted therapy off label.
  Interventions: Drug: CDK4/6 and MEK inhibitor
- C. NRAS mutant melanoma (Experimental): Patients with an NRAS mutation detected on standard gene testing only will receive combined trametinib and ribociclib based on evidence that combining MEK inhibition and CDK4/6 inhibition is a viable treatment option.
  Interventions: Drug: CDK4/6 and MEK inhibitor
- D. BRAF V600 mutant melanoma (Other): Patients will receive standard of care treatment only.
  Interventions: Drug: Standard therapy or clinical trial

INTERVENTIONS:
Drug: Standard therapy or clinical trial — Patients with BRAF V600 mutations detected by standard of care tumour testing will be treated with standard approved therapies or on clinical trials.
  Other Names: Immunotherapy; Biological agent
  Arms: D. BRAF V600 mutant melanoma
Drug: Matched targeted therapy — Patients with tumour found to be non-V600 BRAF, BRAF wildtype and NRAS wildtype melanoma will have tumour tested further using the extended molecular testing platform designed for this project. Patients will first receive standard therapy(ies) for non-V600 BRAF, wildtype and NRAS wildtype melanoma until disease progression or intolerable drug toxicities. Followed by a targeted therapy matched to the genetic aberration detected in their tumour on NGS testing.
  Other Names: ALK - Ceritinib; BRAF fusion - Trametinib; CCND1 - Ribociclib + Trametinib; CDK4/6 - Ribociclib + Trametinib; CDKN2A - Ribociclib + Trametinib; GNA11 - Trametinib; GNAQ - Trametinib; HRAS - Trametinib; KIT - Pazopanib; KRAS - Trametinib; MAP2K1 - Trametinib; NF1 - Trametinib; MET - Ceritinib; RAS - Ribociclib + Trametinib; ROS1 - Ceritinib
  Arms: A1. Non-V600 BRAF, BRAF wildtype, NRAS wildtype. Actionable gene mutation, matched drug available
Drug: Trametinib and / or supportive care — Patients with non-V600 BRAF, BRAF wildtype and NRAS wildtype melanoma for whom there is no actionable genetic aberration found on extended molecular testing, may receive trametinib (if not already administered as part of standard care) and/or supportive care.
  Other Names: Trametinib; Supportive care
  Arms: A3. Non-V600 BRAF, BRAF wild type and NRAS wild type melanoma - no actionable genetic aberration
Drug: CDK4/6 and MEK inhibitor — Patients mucosal melanoma and any genetic aberration on NGS testing may receive ribociclib + trametinib initially. After failure of trametinib and ribociclib, actionable genetic aberrations from the NGS testing will be reviewed for the opportunity to use a further targeted therapy off label.
  Patients with an NRAS mutation on standard of care tumour testing will also receive ribociclib + trametinib.
  Other Names: Ribociclib + Trametinib
  Arms: B. Mucosal melanoma; C. NRAS mutant melanoma
Drug: Compassionate Access Targeted Therapy — Patients with non-V600 BRAF, BRAF wildtype and NRAS wildtype melanoma may have an actionable aberration(s) for which there is no current study-specific drug supply. In this scenario, access will be sought for compassionate use of the off label use of the relevant regulatory approved targeted therapy
  Other Names: Off label use of a matched targeted therapy currently unavailable to the study
  Arms: A2. Non-V600 BRAF, BRAF wildtype, NRAS wildtype. Actionable gene mutation, no matched drug available

SUMMARY:
This is a patient oriented translational research project aiming to improve clinical outcomes for patients with BRAF and NRAS wild-type unresectable Stage III or Stage IV metastatic melanoma who have progressed on, or are unable to receive standard therapy (in general, immunotherapy). Consecutive patients seen at three major clinics and fitting the broad eligibility criteria will be invited to participate.

The approach is designed to test the impact of different targeted drugs on different mutations in a single type of cancer. In this project, patients will have tumour tissue genetically profiled to determine which mutation(s) are present, and will then be assigned to receive a matched drug expected to target the mutation(s) in the tumour. Where multiple targets are identified in one patient, or where multiple potential therapies would be appropriate for a single tumour mutation, the treating clinician may determine the appropriate therapeutic approach after consultation with the study team, using the latest version of library of matched therapies.

DETAILED DESCRIPTION:
Current standard of care testing covers mutations in the BRAF and NRAS genes. The comprehensive gene testing platform to be used in this project is designed to interrogate the entire coding sequence of 315 cancer-related genes plus introns from 28 genes often rearranged or altered in cancer. These genes are known to be somatically altered in solid cancers based on recent scientific and clinical literature. The test panel will be used on melanoma tissue from patients pre-screened as having BRAF and NRAS wild-type melanoma. The extent of testing will be updated to reflect new discoveries in melanoma tumourigenesis and availability of new therapies as the project proceeds. Testing will be performed on formalin-fixed and paraffin-embedded samples of metastatic tissue. Archival tissue from primary or regional recurrent melanoma may be considered if no recent sample is available or possible.

All new patients with unresectable Stage III or IV melanoma seen at each participating site will be invited to participate. Following written consent, all patients will undergo the standard testing for BRAF and NRAS mutations. Patients found to have mutations in either gene will receive standard treatment with dabrafenib and / or trametinib and no further molecular testing.

Patients with wild type versions of BRAF and NRAS genes will have tumour tissue sent for the extended gene testing platform. These patients will first receive standard of care therapy for wild type BRAF / NRAS melanoma, where possible. Once standard therapies have been exhausted (because of disease progression or intolerable adverse events), patients will then receive a targeted therapy matched for their genetic result, if applicable. The selection of targeted therapy will be based on clinical evidence of activity in other solid tumours harbouring similar mutations and / or in at least Phase I testing in melanoma. The table of matched therapies will be modified and extended as new findings from clinical research become available. Patients may be included in specific clinical trials of targeted therapies if available, e.g. a MEK inhibitor combined with an MDM2 inhibitor (AMG232) for BRAF and TP53 wild-type melanoma or a MEK inhibitor combined with a CDK4/6 inhibitor for BRAF wild-type melanoma.

The extensive molecular profiling platform is fully validated and will be conducted by an external provider accredited by an authority with the responsibility to award Laboratory Accreditation at private and public facilities.

ELIGIBILITY:
Inclusion criteria for Part 1:

1. Written informed consent for Part 1
2. Newly diagnosed, histologically confirmedand , unresectable Stage IIIB, IIIC or Stage IV melanoma including cutaneous (including acral, ungual subtypes), ocular (including uveal and extra-uveal), mucosal, and unknown primary).
3. Treatment-naïve for unresectable advanced orf metastatic melanoma (systemic treatment given in the neoadjuvant and adjuvant settings are acceptable).
4. Tumour tissue available from advanced or metastatic disease. Archival tissue from primary or regional recurrent melanoma may be considered if no recent sample is available.
5. Male or female patients aged 18 or over.
6. Standard of care molecular tumour testing which has identified NRAS wild type, and either BRAF wild type or non-V600 BRAF mutant melanoma.
7. Adequate tissue available for the Molecular Testing Platform.

Eligibility Criteria for NGS Molecular Testing Platform (Part 1)

1. Standard of care molecular tumour testing which has identified non V600 BRAF or BRAF wild type, or NRAS wild type melanoma (NRAS mutant patients are eligible for Part 2, but will not undergo NGS testing).
2. Adequate tissue available per NGS specimen preparation instructions.

Inclusion Criteria for Part 2:

1. Written informed consent to receive targeted therapy (if applicable) and clinical follow up.
2. Patient has undergone NGS tumour testing or has NRAS or ALKati mutant melanoma on routine testing
3. Histologically confirmed melanoma of any sub type with measurable disease per RECIST criteria.
4. Received available standard therapies or clinical trial agents for unrectable metastatic melanoma that has progressed, unable to tolerate standard therapy, or standard therapy is contraindicated.
5. Patient has an 'actionable' genetic aberration and matched targeted therapy is available. Patients with no genetic aberration or where no matched targeted therapy is available, patients will be offered trametinib
6. ECOG status 0 - 2.
7. Adequate haematological, hepatic and renal organ function as defined by:

   1. White cell count ≥ 2.0 × 109/L
   2. Neutrophil count ≥ 1.5 × 109/L
   3. Haemoglobin ≥ 90 g/L
   4. Platelet count ≥ 100 x 109/L
   5. Total bilirubin ≤ 3.0 x ULN
   6. Alanine transaminase ≤ 3.0 x ULN
   7. Aspartate aminotransferase ≤ 3.0 x ULN
   8. Serum creatinine ≤ 1.5 x the upper limit of normal (ULN).
8. Life expectancy > 30 days.
9. Women of child bearing potential (WOCBP) to use contraception to avoid pregnancy.
10. Non sterile men with female partners of CBP to use contraception to avoid pregnancy.

Exclusion criteria for Matched Targeted Therapy:

1. An expectation for the need for concurrent radiotherapy (unless safety has been established with the matched drug regimen and is directed at one anatomical region for symptom control).
2. Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug.
3. Any investigational drug or other systemic drug therapy for melanoma within 14 days or 5 half-lives from baseline, whichever is shorter.
4. Pregnant or breast feeding females.
5. Drug specific exclusions as detailed in the TGA Product Information for each drug.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Type and frequency of genetic aberrations in BRAF/NRAS wild-type metastatic melanoma | For the duration of the study, estimated at 5 years.
  Genetic aberrations detected by extended molecular profiling in patients with BRAF / NRAS wild type metastatic melanoma.
Proportion of patients with BRAS/NRAS wild-type melanoma receiving targeted therapy | For the duration of the study, estimated at 5 years.
  Patients able to receive matched targeted therapy as a result of genetic aberrations detected with extended molecular profiling, from a pool of all BRAF / NRAS wild type patients.

SECONDARY OUTCOMES:
Proportion of patients who have BRAF/NRAS wild type melanoma | For the duration of the study, estimated at 5 years.
  From consecutive patients with metastatic melanoma tested for common BRAF / NRAS mutations as part of standard care.
Proportion of patients with complete (CR) or partial (PR) response. | From date of targeted therapy commencement until the date of first documented objective partial or complete response per RECIST, assessed up to 60 months.
  Proportion of patients who received matched targeted therapy as a result of genetic aberrations detected with extended molecular profiling who had a complete (CR) or partial (PR) response.
Duration of response | From date of first objective partial or complete response to disease progression or death, which ever is sooner, assessed up to 60 months.
  For patients experiencing a complete or partial response to study treatment, the amount of time from this outcome to the time that disease progression or death occurs
Progression free survival | From date of targeted therapy commencement to date of objective disease progression per RECIST, assessed up to 60 months.
  The period of time from study entry to progression of disease or death
Overall survival | From date of targeted therapy commencement to date of death from any cause, assessed up to 60 months.
  The proportion of patients alive from the time of study entry
Correlation of genetic aberration detected in tumour tissue with clinical response and disease progression | From date of targeted therapy commencement to date of to partial or complete response or disease progression, assessed up to 60 months.
  Identify genetic predictors of response and progression using the extended molecular testing platform.
Correlation of with genetic aberration detected in tumour tissue with age at diagnosis, site of primary tumour, chronic sun damaged skin. | At baseline
  Identify clinicopathological correlates (e.g. age at diagnosis, site of primary tumour, chronic sun damaged skin etc.) of molecular subtypes of melanoma at baseline.
Correlation of genetic aberration detected in tumour tissue with site of metastases, nodular or superficial spreading disease. | At baseline
  Identify the differences in disease behaviour (e.g. site of metastases, nodular or superficial spreading disease) based on molecular subtypes of melanoma.
Adverse events in patients receiving matched targeted therapy. | From date of the start of targeted therapy to 30 days from discontinuation of targeted therapy
  Characterisation of adverse events by type, frequency and severity using CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Alex Menzies, Study Chair — Melanoma Institute Australia
Locations (2):
- Australia (2):
  - Westmead Hospital, Westmead, New South Wales
  - Melanoma Institute Australia, Wollstonecraft, New South Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nassar KW, Hintzsche JD, Bagby SM, Espinoza V, Langouet-Astrie C, Amato CM, Chimed TS, Fujita M, Robinson W, Tan AC, Schweppe RE. Targeting CDK4/6 Represents a Therapeutic Vulnerability in Acquired BRAF/MEK Inhibitor-Resistant Melanoma. Mol Cancer Ther. 2021 Oct;20(10):2049-2060. doi: 10.1158/1535-7163.MCT-20-1126. Epub 2021 Aug 10. PMID 34376578